CLINICAL TRIAL: NCT04080011
Title: A Case Series Study of Negative Pressure Platform Wound Device (NP-PWD) on the Healing of Elective Surgical Incisions
Brief Title: A Case Series Study of Negative Pressure Platform Wound Device
Acronym: NP-PWD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Metis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-PWD 01
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Incisions, Surgical
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- NP-PWD application (Experimental): All patients enrolled into the study will have the negative pressure- platform wound device applied to their surgical incision.
  Interventions: Device: NP-PWD

INTERVENTIONS:
Device: NP-PWD — Application of NP-PWD device.

SUMMARY:
This primary case series study will demonstrate the safety and feasibility of the NP-PWD technology and treatment protocol to promote healing of surgical incision healing. In a first use in humans of the NP-PWD's capability to deliver negative pressure wound treatment (NPWT), this project will gather data from patients with elective surgical incisions, with the intention to evaluate the NPWT capability for future use in more tenuous situations of wound closure.

DETAILED DESCRIPTION:
A case series study of 10 subjects will be conducted by enrolling patients who are scheduled for elective surgical incisions. Patients will be screened for inclusion criteria and asked to consent to participate in the study for single application treatment with the NP-PWD for 3-6 days. Initial evaluation of the incision would occur on Day 0, including screening, pre-procedure evaluation, measurement and photography of the closed surgical incision. Follow up data is then gathered Day 3-6 with removal of the NP-PWD, surgical incision assessment and photography, and assessment for adverse effects. Day 9-14 follow up include the same assessments of progression of wound closure. Gathered clinical data of the 10 subjects will be used to evaluate the safety in using the NPWT device for effective wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-85 years of age.
2. Scheduled for surgical intervention in which an incision will be made and skin closure will be performed.

Exclusion Criteria:

1. Active infection as judged by the Investigator
2. Inability to give informed consent
3. Active malignant disease or subject is less than one year disease-free
4. Use of immunosuppressive agents, radiation or chemotherapy within the past 30 days
5. Any concomitant medications or co-morbidities that, in the opinion of the investigator, may interfere with wound healing
6. On any investigational drug(s) or therapeutic device(s) in the last 30 days or any previous enrollment in this study
7. Pregnant at enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events. | Three to six days post application.
  Safety is assessed by recording each adverse event (AE) occurring during the period the patient has the study device applied and throughout the entire enrollment period.
Rate of successful application of the NP-PWD device | Three to fourteen days post application
  Descriptive data collected: device application, device removal, adverse device effects, device errors, device complications, and resultant in healing status of the surgical incision.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events. | Fourteen days post application.
  Safety is assessed by recording each adverse event (AE) occurring during the period the patient has the study device applied and throughout the entire enrollment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Northeast Baptist, San Antonio, Texas, United States